CLINICAL TRIAL: NCT00189943
Title: Phase I Study on Safety, Tolerability and Immunogenicity of the MVA-BN Vaccine Administered to Healthy Subjects
Brief Title: Study on Safety, Tolerability and Immunogenicity of an MVA Vaccine Administered to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MVA-POX-001; Bavarian Nordic
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2005-09-19 (Estimated); Status verified 2005-09

CONDITIONS: Smallpox
MeSH Terms: conditions — Smallpox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

INTERVENTIONS:
Biological: MVA-BN

SUMMARY:
The purpose of this study is to collect information on the safety, tolerability and immunogenicity of an investigational smallpox vaccine at different doses and using different routes of administration in vaccinia-naive and vaccinated healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, aged 20 - 55 years
* Signed informed consent

Exclusion Criteria:

* Prior vaccination against smallpox (study part I only)
* Abnormalities suspicious of any underlying disease, detected at routine tests prior to study inclusion.
* Any immune modifying therapy within 4 weeks prior to entry
* Participation in any other investigating drug trial
* Known allergy to a component which may be part of the vaccine
* Allergic reaction or any other severe adverse effects experienced after previous smallpox vaccination (study Part II only)

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90
Dates: Start 2001-04; Study Completion 2003-07

CONTACTS AND LOCATIONS:
Overall Officials: Karl M Eckl, MD, Principal Investigator — PharmPlanNet Cantract Research GmbH
Locations (1):
- PharmPlanNet Contract Research GmbH, Mönchengladbach, Germany